CLINICAL TRIAL: NCT06737731
Title: A Phase I/II, Multicenter, Open-Label Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-1681 for Injection in Patients With Malignant Solid Tumors
Brief Title: A Phase I/II Clinical Study of SHR-1681 for Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1681-101
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1681 (Experimental)
  Interventions: Drug: SHR-1681

INTERVENTIONS:
Drug: SHR-1681 — SHR-1681 for Injection will be administrated per dose level in which the patients are assigned.

SUMMARY:
This study is an open-label, multicenter Phase I/II clinical trial to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-1681 for injection in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form;
2. Subjects with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors which is relapsed or refractory to standard treatment, or lack of standard treatment, or standard treatment is not applicable currently;
3. Have at least one measurable tumor lesion per RECIST v1.1;
4. ECOG performance score of 0-1;
5. Life expectancy ≥ 3 months;
6. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Subjects with active central nervous system metastases or meningeal metastases;
2. History of serious cardiovascular and cerebrovascular diseases;
3. Subjects with a history of interstitial pneumonitis or imaging at screening suggestive of suspected interstitial pneumonitis;
4. Severe infection within 4 weeks prior to the first dose;
5. Ongoing or previous anti-tumor therapies within 4 weeks prior to the first dose of study drug;
6. Adverse reactions of previous anti-tumor treatment have not recovered to Grade ≤ 1 per NCI-CTCAE v5.0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 12 months.
Maximum administered dose (MAD) | 12 months.
Recommended Phase 2 dose (RP2D) | 12 months.
Incidence and severity of adverse events (AEs) | Approximately 3 years.
Incidence and severity of serious adverse events (SAEs) | Approximately 3 years.

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of SHR-1681 | Approximately 3 years.
Maximum concentration (Cmax) of SHR-1681 | Approximately 3 years.
Area under the concentration-time curve from time 0 to the last measurable concentration time point (AUC0-t) of SHR-1681 | Approximately 3 years.
Area under the concentration-time curve from time 0 to infinity (AUC0-∞) of SHR-1681 | Approximately 3 years.
Anti-SHR-1681 antibody (ADA) of SHR-1681 | Approximately 3 years.
Overall response rate (ORR) | Approximately 3 years.
Duration of response (DoR) | Approximately 3 years.
Disease control rate (DCR) | Approximately 3 years.
Progression-free survival (PFS) | Approximately 3 years.
Overall survival (OS) | Approximately up to 5 years after the last subject enrolled.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Dongfang Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided